CLINICAL TRIAL: NCT06514755
Title: Sequential Genicular Nerve Ablation Prior to Geniculate Artery Embolization in Knee Pain Management: A Randomized Controlled Trial
Brief Title: Sequential Genicular Nerve Ablation Prior to Geniculate Artery Embolization in Knee Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Awad Bessar, Assistant Professor of Diagnostic and Interventional Radiology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GNA-GAE-KP
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Chronic Knee Pain; Osteoarthritis
Keywords: Genicular Nerve Ablation; Geniculate Artery Embolization; Knee Function; Patient Satisfaction
MeSH Terms: conditions — Osteoarthritis; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: one undergoing sequential genicular nerve ablation (GNA) followed by geniculate artery embolization (GAE), and the other receiving GAE alone.
Who Masked: Outcomes Assessor
Masking Description: Given the specific nature of the interventions, it may not be possible to blind participants or operators; however, to minimize potential bias, outcome assessors will be blinded to the treatment assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential GNA Followed by GAE (Experimental): Participants in this group will undergo genicular nerve ablation (GNA), followed by geniculate artery embolization (GAE) one month later. The GNA procedure will target the genicular nerves responsible for knee pain, and the GAE procedure will target the geniculate arteries to reduce inflammation and pain. The sequence is designed to optimize pain relief and functional outcomes.
  Interventions: Procedure: GNA followed by GAE
- GAE Alone (Active Comparator): Participants in this group will receive geniculate artery embolization (GAE) alone, without prior genicular nerve ablation (GNA). The GAE procedure will target the geniculate arteries to reduce inflammation and pain. This arm serves as the control to compare the effectiveness and safety of the sequential GNA followed by GAE intervention.
  Interventions: Procedure: GAE alone

INTERVENTIONS:
Procedure: GNA followed by GAE — Participants in the experimental arm will undergo genicular nerve ablation (GNA), a minimally invasive procedure targeting the genicular nerves to interrupt pain transmission. One month after undergoing GNA, participants will receive geniculate artery embolization (GAE), which targets the geniculate arteries to reduce inflammation and pain.
  Arms: Sequential GNA Followed by GAE
Procedure: GAE alone — Participants in the active comparator arm will receive geniculate artery embolization (GAE) alone, a minimally invasive procedure targeting the geniculate arteries to reduce inflammation and pain, without prior genicular nerve ablation (GNA).
  Arms: GAE Alone

SUMMARY:
The goal of this clinical trial is to evaluate whether performing genicular nerve ablation (GNA) before geniculate artery embolization (GAE) improves pain relief and knee function in patients with chronic knee pain. The main questions it aims to answer are:

* Does performing GNA prior to GAE enhance pain relief, as measured by the Visual Analog Scale (VAS), at 3 months post-procedure?
* Does the sequential approach improve knee function as assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)?

Study investigators will compare two groups to see if the sequential approach (GNA followed by GAE) provides better outcomes compared to GAE alone.

Participants will:

* Undergo either sequential GNA followed by GAE or GAE alone
* Have their knee pain and function assessed at baseline, 1 month, 3 months, and 6 months post-procedure
* Complete a structured patient satisfaction questionnaire (PSQ) at 3 months post-procedure
* Be monitored for procedure-related adverse events up to 6 months post-procedure,

DETAILED DESCRIPTION:
Background:

Chronic knee pain is a prevalent condition affecting a significant portion of the population, often leading to reduced quality of life and functional impairment. Current treatment options include genicular nerve ablation (GNA) and geniculate artery embolization (GAE). However, the optimal sequence of these interventions remains unclear.

Rationale:

The rationale for investigating the sequence of genicular nerve ablation (GNA) followed by geniculate artery embolization (GAE) lies in potentially optimizing pain relief and functional outcomes while ensuring patient safety and satisfaction. GNA aims to interrupt pain transmission from the genicular nerves to the central nervous system, while GAE targets the blood supply to the inflamed synovium, reducing inflammation and pain. Understanding whether performing GNA prior to GAE offers superior pain relief, functional improvement, and patient satisfaction compared to GAE alone is crucial for optimizing treatment protocols and guiding clinical practice.

Objectives:

1. Primary Objective:

   - Evaluate whether performing GNA prior to GAE enhances pain relief, as measured by the Visual Analog Scale (VAS), at 3 months post-procedure.
2. Secondary Objectives:

   * Evaluate changes in knee function using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), a validated scoring system specifically designed for osteoarthritis.
   * Monitor and document any procedure-related adverse events to compare the safety profiles of both techniques.
   * Evaluate patient satisfaction using the structured Patient Satisfaction Questionnaire (PSQ).

Study Design:

This study is a randomized controlled trial (RCT) aimed at evaluating the effectiveness of sequential GNA followed by GAE versus GAE alone in managing chronic knee pain. Eligible patients will be randomly allocated to one of the two treatment groups. Given the specific nature of the interventions, it may not be possible to blind participants or operators; however, to minimize potential bias, outcome assessors will be blinded to the treatment assignments.

Interventions:

1. Sequential Genicular Nerve Ablation (GNA) followed by Geniculate Artery Embolization (GAE): Participants will undergo GNA targeting genicular nerves followed by GAE targeting geniculate arteries. Ablation parameters and embolization procedures will be standardized to ensure consistency across interventions.
2. Geniculate Artery Embolization (GAE) Alone: Participants assigned to this group will receive GAE without prior GNA. The embolization procedure will follow standard protocols to target the geniculate arteries effectively.

Outcomes:

a) Primary Outcome

- Reduction in Knee Pain; this measure assesses the change in knee pain as reported by participants using the Visual Analog Scale (VAS). A lower score indicates less pain, signifying an improvement.

Secondary Outcomes:

* Improvement in Knee Function; Assessed by changes in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores, which measure pain, stiffness, and physical function of the knee and hip joints. A lower WOMAC score indicates better joint function.
* Incidence of Procedure-Related Adverse Events; monitoring and recording any adverse events related to the genicular nerve ablation procedures.
* Patient Satisfaction with the Procedure; measured using a structured patient satisfaction questionnaire (PSQ) to gauge participants' satisfaction with the pain relief and overall experience of the procedure.

Follow-Up: Participants will be closely monitored post-procedure with scheduled follow-up visits at 1 week, 1 month, 3 months, and 6 months. These visits will include clinical assessments, pain evaluations, functional tests, and documentation of any adverse events.

Conclusion: This study aims to provide valuable insights into the effectiveness, safety, and patient satisfaction of performing genicular nerve ablation prior to geniculate artery embolization in the management of chronic knee pain. By rigorously evaluating these techniques, the findings will inform clinical decision-making, optimize treatment strategies, and pave the way for future research aimed at enhancing outcomes for patients suffering from chronic knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years.
* Diagnosed with chronic knee pain refractory to conservative treatment.
* Able to provide informed consent.
* Agree to follow the study procedures and attend follow-up visits.

Exclusion Criteria:

* Contraindications to GNA or GAE procedures (e.g., allergy to local anesthetics, active infection at the procedure site).
* Recent knee surgery within the last six months.
* Severe comorbid conditions that may interfere with the study outcomes (e.g., rheumatoid arthritis, other severe autoimmune diseases).
* Current participation in another clinical trial that could interfere with the outcomes of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Knee Pain | 3 months post-procedure
  This outcome measures the change in knee pain as reported by participants using the Visual Analog Scale (VAS). A lower score indicates less pain, signifying an improvement.

SECONDARY OUTCOMES:
Improvement in Knee Function | Assessed at 1 month, 3 months, and 6 months post-procedure
  Assessed by changes in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores, which measure pain, stiffness, and physical function of the knee and hip joints. A lower WOMAC score indicates better joint function.
Incidence of Procedure-Related Adverse Events | From the time of procedure up to 6 months
  Monitoring and recording any adverse events related to the genicular nerve ablation procedures
Patient Satisfaction with the Procedure | 3 months post-procedure
  Measured using a structured patient satisfaction questionnaire (PSQ) to gauge participants' satisfaction with the pain relief and overall experience of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Bessar, MD, PhD, Principal Investigator — Assistant Professor of Diagnostic and Interventional Radiology, Zagazig Uni.
Locations (1):
- Zagazig University, Faculty of Medicine, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) with other researchers. This decision is based on considerations related to patient confidentiality, data privacy concerns, and the absence of a current infrastructure for secure data sharing. The primary results of the study will be published in peer-reviewed journals and presented at scientific conferences, ensuring that the findings are accessible to the broader research community.